CLINICAL TRIAL: NCT06731244
Title: Prognosis Improvement of Unprovoked vEnous THromboEmbolism With the Use of a Shared Decision-making Process Including a Time-dependent Multicomponent Risk Prediction Scores inteRvention.
Brief Title: Shared Decision-making Process for Unprovoked vEnous THromboEmbolism Management. (ETHER )
Acronym: ETHER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: European Commission (Other); European Clinical Research Infrastructure Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 29BRC23.0189; 2024-A01652-45 (Other: IDRCB)
Record Dates: First submitted 2024-11-08; First posted 2024-12-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Venous Thromboembolism
Keywords: venous thrombosis; pulmonary embolism; Anticoagulant; deep vein thrombosis; stepped-wedge cluster randomized trial; shared-decision making
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: ETHER is a stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Anticoagulant treatment management according to usual practice and international guidelines
  Interventions: Other: Usual Care Group
- Experimental arm (Experimental): Shared decision-making process integrating time-dependent multicomponent risk prediction scores and socio-anthropological scales (TDMI)
  Interventions: Other: shared decision-making process

INTERVENTIONS:
Other: Usual Care Group — Patients will be managed as regards their anticoagulant treatment according to usual practice and in accordance with international guidelines.
  Arms: Control arm
Other: shared decision-making process — The intervention is based on a strategy based on a shared decision-making process which is a collaborative process that involves a patient and their healthcare professional working together to reach a joint decision about care (anticoagulant treatment).
  The shared decision-making process will be conducted as follows:
  * Step 1: prepare the risk estimates (risk of recurrent VTE, risk of bleeding) for the patient, based on time-dependent multicomponent risk prediction scores and socio-anthropological scales (TDMI) and other validated risk prediction scores and evidence-based medicine;
  * Step 2: Communicating risks, benefits and consequences to the patient;
  * Step 3: Make a joint decision about treatment and care, and agree together when this will be reviewed.
  Arms: Experimental arm

SUMMARY:
Venous thromboembolism (VTE) including deep vein thrombosis (DVT) and pulmonary embolism (PE) is a frequent disease and the third most common cause of cardiovascular death in the world after myocardial infarction and stroke. Anticoagulant therapy drastically reduces the risk of early VTE recurrence and death, but it exposes patients to a substantial risk of bleeding. Hence, determining the optimal duration of anticoagulant treatment for VTE is a major public health issue.

When major transient risk factors for VTE are identified (major surgery, immobilization...), patients generally do not need to extend anticoagulation beyond 3 months, whereas for VTE diagnosed in the context of cancer, therapeutic anticoagulation is required for as long as the cancer is considered "active".

However, in more than 50% of cases, venous thromboembolic disease occurs spontaneously, i.e. without any significant clinically detectable circumstance (known as unprovoked venous thromboembolic disease). In such patients, the risk of recurrence is high (35% recurrence rate at 5 years, with a 10% risk of death per recurrence). Scientific societies therefore recommend continuing anticoagulant treatment "indefinitely" (i.e. without programming a stop date or long-term treatment). However, this practice exposes these patients to an ongoing, non-negligible increase in the risk of bleeding, which could ultimately exceed the risk of recurrence of venous thrombo-embolic disease.

Optimizing anticoagulant therapy beyond the first three to six months of treatment is therefore a crucial and challenging issue, which could improve the long-term prognosis of patients with unprovoked thromboembolic venous disease.

Based on the quantitative and qualitative approaches implemented in MORPHEUS project granted by European Commission (HORIZON-HLTH-2022-TOOL-11-01 call), the investigators have combined predictive personalized medicine, through the use of risk biomarkers, with a patient-centered model of medicine, which, while based on an understanding of the patient's experience, leading to develop Time-Dependent Multicomponent risk prediction scores and socIo-anthropological scales (TDMI) integrated in a shared decision-making process regarding anticoagulant treatment duration in patients with a first episode of unprovoked VTE.

The aim of this study is to demonstrate that this strategy, based on a medical decision-making process shared between patients and physicians and including TDMI, reduces the risk of recurrence of thromboembolic venous disease (fatal or non-fatal), the risk of bleeding and all-cause mortality, and is associated with greater patient satisfaction after a first episode of unprovoked thromboembolic venous disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient > or = 18 years,
* Patient with a first episode of symptomatic unprovoked pulmonary embolism (PE) and/or proximal deep vein thrombosis (DVT) treated for 3 to 6 uninterrupted months with full dose anticoagulant therapy,
* Signed informed consent.

Exclusion Criteria:

* Unable or refusal to give informed consent,
* Isolated distal DVT,
* Isolated sub-segmental PE
* Previous unprovoked VTE
* Known CTEPH
* Indication for anticoagulation other than DVT or PE (e.g.; atrial fibrillation, mechanic valves…),
* Interruption of anticoagulation for 14 days or more before the inclusion,
* Active cancer of less than 24 months,
* Current pregnancy,
* Life expectancy <18 months (e.g.; patients with an end-stage chronic disease)
* Not affiliated to national insurance, social security (only for France)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2035-10 (Estimated); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite of adjudicated all-cause mortality, adjudicated symptomatic recurrent VTE (fatal or non-fatal PE or proximal DVT), adjudicated major and clinically relevant non-major bleeding, and patient's satisfaction | From inclusion to 18th month follow-up
  For the statistical analysis, the investigators will analyse hierarchically each component of the composite (all-cause mortality, then VTE recurrence, then major bleeding or clinically relevant non-major bleeding and then patient's satisfaction in this order) using a win ratio approach to assess the primary composite outcome.

SECONDARY OUTCOMES:
Composite of adjudicated all-cause mortality, symptomatic recurrent VTE (fatal or non-fatal PE or proximal DVT) and major and clinically relevant non-major bleeding | At 18-month follow-up after inclusion
  This clinical composite outcome will be compared between the intervention group and the control group at the individual level with a mixed effect cox model with a random intercept to account for the correlation between patients of a same cluster. The random intercept will correspond to a random period effect nested in a random cluster effect. Different covariance structure will be tested, the model will be selected as the best identifiable model that produces the lowest Bayesian Information Criterion (BIC) value. The effect of the intervention (shared decision-making process including a TDMI) will be then presented as the hazard ratio between the two groups of treatment and its corresponding 95% CI. A random cluster effect will be added to the treatment group effect, if necessary, to quantify any heterogeneity in the benefit of the intervention. The superiority test on this outcome will be performed only if the primary outcome is statistically demonstrated.
Adjudicated all-cause mortality, | At 18 months follow-up after inclusion
Adjudicated symptomatic VTE recurrence | At 18-month follow-up after inclusion
Adjudicated major bleeding or clinically relevant non-major bleeding | At 18-month follow-up after inclusion
Adjudicated fatal recurrent VTE and fatal bleeding | At 18-month follow-up after inclusion
Patient's satisfaction | At 18-month follow-up after inclusion
  Patient's satisfaction will be defined with the Patient Activation Measure - PAM score using 13 items measures that assess patient's knowledge, skill, and confidence for self-management. The scoring (for each criteria) is:
  * Strongly disagree = 1
  * Disagree = 2
  * Agree = 3
  * Strongly agree = 4
Quality of life (QoL) assessed using PembQoL questionnaire | At 18 months after inclusion
  Evaluation only for patients with symptomatic PE. The PEmb-QoL Score is ranged between 0% and 100% for each of its 6 dimensions. Higher scores indicate worse outcome.
Quality of life (QoL) assessed using mMRC dyspnea score | At 18 months after inclusion
  Evaluation only for patients with symptomatic PE. Scale ranged from 0 (no dyspnea) to 5 (worst grade)
Quality of life (QoL) assessed using VEINQol questionnaire | At 18 months after inclusion
  Evaluation only for patients with symptomatic DVT. Responses are rated on two-point to seven-point Likert response scales of intensity, frequency, or agreement.
Quality of life (QoL) assessed using Villalta score | At 18 months after inclusion
  Evaluation only for patients with symptomatic DVT. The total Villalta score, ranging from 0 to 33, will be assessed in both legs and used to categorize the severity of PTS in the index leg as mild (score, 5-9), moderate (score, 10-14), or severe (score, ≥15 or presence of ulceration).
Quality of life (QoL) assessed using EQ-5D5L questionnaire | At 18 months after inclusion
  Five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels. The patient is asked to indicate his/her health state.
Quality of life (QoL) assessed using PVFS scale patients | At 18 months after inclusion
  Scale ranged from 0 (normal functional status) to 5 (worse grade)
Therapeutic adherence to anticoagulant treatment | At18-month follow-up after inclusion
  Therapeutic adherence using Girerd's questionnaire: 6 items. Score 0 = good compljance ; Score 1-2 = minor concern in compliance ; Score ≥ 3 = bad compliance.
Occurence of objectively diagnosed cancer: site, localized, locally advanced, metastatic | From inclusion to 18th months follow-up
  Cancers will be classified according the site and the extend (localized, locally advanced, metastatic).
Occurence of minor or atypical venous thrombosis | At 18-month follow-up after inclusion
  Minor venous thrombosis includes superficial vein thrombosis, muscular and distal deep vein thrombosis. Atypical venous thrombosis includes: Proximal upper limbs Superior vena cava, Cerebral venous thrombosis, Portal thrombosis, Mesenteric thrombosis, Sus-hepatic vein thrombosis, Renal thrombosis, Ovarian vein thrombosis, Uterine vein thrombosis, Retinal vein thrombosis.
Adjudicated objectively diagnosed acute arterial thromboembolic events according to international guidelines: stroke, myocardial infarction, peripheral arterial thromboembolic event, atrial fibrillation, any cardiac event other than VTE | At 18-month follow-up after inclusion
Adjudicated objectively confirmed chronic thromboembolic pulmonary disease and chronic thromboembolic pulmonary hypertension | At 18-month follow-up after inclusion

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU Brest, Brest, France
  - CHU d'Amiens - Picardie, Amiens
  - CHU d'Angers, Angers
  - Hôpital National d'Instruction des Armées Percy, Clamart
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - APHP-Colombes, Colombes
  - CHU de Dijon - Hôpital François Mitterand, Dijon
  - CH Le Mans, Le Mans
  - HCL - Hôpital Edouard Herriot, Lyon
  - APHM - Hôpital la Timone, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - Aphp-Hegp, Paris
  - CHU de Rennes, Rennes
  - CHU Saint Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse